CLINICAL TRIAL: NCT06920927
Title: Feasibility and Pilot Testing of the "My Heart and CKD" Online Shared Decision Aid
Brief Title: Feasibility and Pilot Testing of "My Heart and CKD" Online Shared Decision Aid
Acronym: MyHeart&CKD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of Alberta (Other); Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: REB22-0289
Record Dates: First submitted 2025-03-11; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease; Coronary Artery Disease
Keywords: Decision aid; Shared decision making
MeSH Terms: conditions — Renal Insufficiency, Chronic; Coronary Artery Disease | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: Cluster randomized stepped wedge design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Decision aid intervention (Experimental): Patients in this group will receive care from their physician incorporating the use of the decision aid.
  Interventions: Other: Decision aid
- Usual Care (No Intervention): Patients in this group will receive usual care from their physician without the use of the decision aid.

INTERVENTIONS:
Other: Decision aid — Decision aid for use by physicians and patients with CKD when deciding upon an invasive vs a conservative approach to management of coronary artery disease.
  Arms: Decision aid intervention

SUMMARY:
Many people with kidney disease also have heart disease. The procedures used to diagnose and treat heart disease (e.g., angiograms, angioplasty, or surgery) can improve symptoms and cardiovascular outcomes, but pose greater risks of kidney complications for people with chronic kidney disease. It's therefore important that patients with kidney disease and their health care providers understand the benefits versus risks of these procedures and use that information to make informed decisions regarding their health care.

Prior research done with patients with kidney disease and their health care providers has led to the develop of a decision aid designed to help doctors provide personalized information on the benefits versus risks of having a heart procedure, as well as help patients communicate their own values and preferences to their doctor. This information is crucial for shared decision making, as previous research has shown that preferences and values vary for individual patients with kidney diseases, and should be incorporated into the decision-making process for heart disease management. The decision aid, called "My Heart Care and CKD", supports shared decision-making between patients with kidney disease and heart their care providers. This trial will implement and evaluate this decision aid within cardiovascular care in a pilot trial in Canada.

DETAILED DESCRIPTION:
Heart disease is a common comorbidity in individuals with chronic kidney disease (CKD). However, patients with CKD are 20-50% less likely to receive heart tests and treatments for acute coronary syndromes and there is also substantial variability in management for patient with CKD and stable coronary disease. The variability and disparities in care for people with CKD are attributed to three common obstacles: concern over potential kidney function deterioration from procedures, limited understanding of the benefits and risks of invasive versus medical treatment approaches for individual patients with CKD, and inadequate strategies to align treatment decisions with patient values and preferences. Addressing these barriers necessitates a shift towards patient-centered care and informed decision-making in cardiovascular and kidney care. Offering personalized risk information and decision support to patients with CKD and their care providers could help surmount these obstacles. These patient-oriented approaches to heart disease care require weighing treatment decisions' risks and benefits through informed discussions between patients and providers.

Shared decision-making (SDM), a collaborative approach between patients and healthcare providers, integrates clinical knowledge with patient values, preferences, and risk tolerance to personalize care decisions. SDM, when integrated into care practices, enhances patient satisfaction and experiences. However, despite its benefits, only a minority of Canadian patients report experiencing SDM, highlighting the need for its broader implementation.

Patient decision aids (PDAs) are tools for facilitating collaborative medical decisions, particularly when multiple treatment options exist. PDAs equip patients with information on treatment choices, associated risks, and benefits, and help them clarify their values in the decision-making process. A Cochrane Systematic Review highlighted that when utilized, PDAs enhance patient knowledge, ensure informed decision-making, and foster active patient involvement in the decision process. Guideline frameworks like the International Patient Decision Aid Standards (IPDAS) and Ottawa Framework ensure the rigor and standardization of PDA development.

Trial Objectives:

This study will implement and evaluate a decision aid for use by patients with CKD and heart disease and their healthcare providers when making treatment decisions for coronary artery disease, including with acute coronary syndrome and stable coronary artery disease.

Specific objectives are:

1. To measure the effectiveness of delivery of personalized information for patients with CKD and heart disease and their health care providers within clinical care. The investigators will measure use and completion of the decision-aid during clinical care encounters for management of heart disease within an implementation pilot trial. Quantitative and qualitative methods will be used to measure how effectively the decision aid conveys personalized information. The investigators will also examine how closely management decisions correlate with risk estimates for patients who received the decision aid. Measures from patients with and without use of the decision aid will be compared using a cluster randomized, pre- versus post-implementation, design, to evaluate effectiveness.
2. To work towards better recognition of patient preferences and their incorporation into decision making, the investigators will measure the knowledge, experience, and satisfaction of patients who receive the decision-aid within the implementation pilot trial. The investigators will compare the expressed preferences of patients to the management approach that patients received and determine whether greater concordance is achieved using the decision aid than observed in the absence of a decision aid.
3. To examine the decision aid's effects on awareness, understanding, and incorporation of shared decision-making practices, the investigators will survey and interview health care providers on knowledge and confidence with shared decision-making before and after use of the decision aid. The investigators will also measure the decisional conflict of patients who received the decision aid and those who did not, which is an outcome measure that has been shown to improve with interventions that support shared decision-making.

Primary objective: Conduct an implementation pilot study in Canada, deploying the decision aid accompanied by implementation training and resources for culturally sensitive shared decision-making within clinical care.

Secondary objective: To document and evaluate the feasibility, acceptability, and satisfaction with use of the decision aid.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age or older)
* Chronic kidney disease
* Coronary artery disease (non-ST elevation acute coronary syndrome (ACS) or symptoms or signs of stable coronary heart disease)
* Able to communicate in English or French or through a support person who speaks English or French
* Patient has the cognitive ability or has a surrogate decision maker capable of participating in shared decision making based on the discretion of the attending physician

Exclusion Criteria:

* End stage kidney failure already being treated with dialysis or with an eGFR < 10mL/min/1.73m2
* ST-elevation myocardial infarction
* Patient is not expected to survive to hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict Scale (O'Connor -8 question) | Following patient-physician encounter (within 2 weeks)
  Patient's perceptions of modifiable factors contributing to uncertainty with their decision such as feeling uninformed, unclear about personal values and unsupported in decision making; and effective decision making such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice.
Patient Nine-item Shared Decision-Making Questionnaire (SDM-Q-9) | Following patient-physician encounter (within 2 weeks)
  Assessment of patient's perceived level of involvement in decision-making related to their own treatment.
Knowledge of Treatment Risks | Following patient-physician encounter (within 2 weeks)
  Patient's knowledge of the risks of kidney failure versus a heart attack in the future associated with the treatment choices of invasive versus optimal medical management presented in the decision aid
Accuracy of Risk Perception | Following patient-physician encounter (within 2 weeks)
  Whether a patient's perception of risk of the risk of kidney failure corresponds to the estimated risk of this outcome for a similar person receiving invasive management as presented in the decision aid
Value-Choice Congruence | Following patient-physician encounter (within 2 weeks)
  Whether a patient's choice of invasive versus optimal medical management is consistent with their most important stated values

SECONDARY OUTCOMES:
Preferred Choice | Following patient physician encounter (within 2 weeks) and 3 months later
  The patient's inclination towards a preferred choice of treatment with invasive versus conservative management
Actual Choice | Following patient-physician encounter (within 2 weeks)
  Whether invasive or optimal medical therapy was actually chosen by the patient and physician.
Adherence to Chosen Option | Three months following the patient-physician encounter
  Whether the treatment received (invasive or medical therapy) remained the same as the initially chosen option
Decisional Regret Scale (O-Connor - 5 question) | Three months following the patient-physician encounter
  Evaluation of feelings of dissatisfaction or disappointment following the decision, reflecting on whether the individual would make the same decision given the chance again
Acceptability Scale (O'Connor - 10 question) | Following patient-physician encounter (within 2 weeks)
  Patient's rating of the comprehensibility of components of a decision aid, its length, amount of information, balance in presentation of information about options, and overall suitability for decision making.
Physician Nine-item Shared Decision-Making Questionnaire (SDM-Q-9) | Following patient-physician encounter (within 2 weeks)
  Assessment of physician's perceived level of patient involvement in decision-making related to their own treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T James, MD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No
Maintenance of data privacy and security .

REFERENCES:
- [Background] Wilson T, Javaheri P, Finlay J, Hazlewood G, Wilton SB, Sajobi T, Levin A, Pearson W, Connolly C, James MT. Treatment Preferences for Cardiac Procedures of Patients With Chronic Kidney Disease in Acute Coronary Syndrome: Design and Pilot Testing of a Discrete Choice Experiment. Can J Kidney Health Dis. 2021 Jan 27;8:2054358120985375. doi: 10.1177/2054358120985375. eCollection 2021. PMID 33552527
- [Background] Finlay J, Wilson T, Javaheri PA, Pearson W, Connolly C, Elliott MJ, Graham MM, Norris CM, Wilton SB, James MT. Patient and physician perspectives on shared decision-making for coronary procedures in people with chronic kidney disease: a patient-oriented qualitative study. CMAJ Open. 2020 Dec 10;8(4):E860-E868. doi: 10.9778/cmajo.20200039. Print 2020 Oct-Dec. PMID 33303572
- [Background] Wilson TA, Hazlewood GS, Sajobi TT, Wilton SB, Pearson WE, Connolly C, Javaheri PA, Finlay JL, Levin A, Graham MM, Tonelli M, James MT. Preferences of Patients With Chronic Kidney Disease for Invasive Versus Conservative Treatment of Acute Coronary Syndrome: A Discrete Choice Experiment. J Am Heart Assoc. 2023 Mar 21;12(6):e028492. doi: 10.1161/JAHA.122.028492. Epub 2023 Mar 9. PMID 36892063
- See also: Shared Decision-Making for Heart and Kidney Disease — https://cansolveckd.ca/research-projects/shared-decision-making-for-heart-and-kidney-disease/